CLINICAL TRIAL: NCT06847893
Title: The Effect of Rebozo Technique on Perceived Support and Control in Childbirth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Collaborators: Uskudar University (Other)
Responsible Party: Principal Investigator, Ayça Demir Yıldırım, PhD, Doctor Faculty Member, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Ü.Ü. Ebe Büşra Ata
Record Dates: First submitted 2025-02-08; First posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Pregnant Women
Keywords: rebozo; support; control; pregnant; birth

STUDY DESIGN:
Intervention Model Description: The study was designed as a randomized controlled, 2-group (intervention and control), experimental research.
Who Masked: Participant
Masking Description: The numbers from 1 to 44 were randomly divided into two groups on the random.org website and randomly selected numbers were assigned to the intervention and control groups. This process ensured equal and random distribution of participants to the intervention and control groups. The group to which the case was assigned was determined according to the order of hospitalization and recorded in the Excel list.
  Since the care intervention and data collection were performed by the researcher in the study, one-way blinding was performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): After the randomization of the women placed in the clinic, they were informed about the study and their consent was obtained; then the Introductory Information Form was completed. The experimental group (n=22) received massage with rebozo technique during the active phase of labor in addition to routine care in accordance with clinical procedures. A 'Rebozo Application Calendar' was created for the experimental group. According to this calendar, 4 rebozo techniques were determined. The duration and frequency of the techniques and the cervical dilatation of the pregnant woman at the time of application were recorded. After delivery, the 'Perceived Support and Control in Childbirth Scale' was completed.
  Translated with DeepL.com (free version)
  Interventions: Other: rebozo technique
- control group (No Intervention): After the randomization of the women placed in the clinic, they were informed about the study and their consent was obtained; then the Introductory Information Form was completed. The control group (n=22) received routine midwifery care only in accordance with clinical procedures. A 'Rebozo Implementation Schedule' was created for the participants in the experimental group. According to this schedule, rebozo techniques to be applied in the latent and active phase of labor were determined. The duration and frequency of the rebozo techniques and the cervical dilatation of the pregnant woman when the technique was applied were recorded. After delivery, the 'Perceived Support and Control in Labor Scale' was completed.

INTERVENTIONS:
Other: rebozo technique — In accordance with the 'Rebozo Chart' developed by the researcher, the pregnant women in the experimental group were massaged with 4 different rebozo techniques (rebozo technique in hand-knee position, rebozo technique in knee-chest position, umbilical support with rebozo, rebozo technique applied with Pilates ball) in the active phase of labor. After the application, the duration, frequency and cervical dilatation of the pregnant woman were recorded in the chart.
  Arms: Experimental Group

SUMMARY:
This study was designed as a randomized controlled, 2-group, experimental study to measure the levels of perceived birth support and control between women with and without rebozo technique.

DETAILED DESCRIPTION:
Objective: This study was conducted to measure the perceived support during labor and the level of control over their own labor in pregnant women who underwent rebozo technique.

Method: The study was conducted in a randomized controlled experimental design between September and December 2024. The population of the study consisted of 44 primiparous pregnant women admitted to a district state hospital for delivery. The sample size was calculated and the study was conducted with 44 pregnant women (experiment: 22, control: 22). While rebozo technique was applied to the experimental group during the trauma process, routine midwifery care was applied to the control group. Introductory Information Form, Perceived Support and Control Scale in Childbirth were used to collect data in the study.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the research,
* Don't speak Turkish,
* Being literate,
* Having a low-risk pregnancy,
* Primiparous pregnancy

Exclusion Criteria:

* Being out of position
* Having a high-risk pregnancy (vaginal bleeding, no hypertension, etc.),
* Dilatation below 4 cm and above 6 cm,
* Initiation of labor induction,
* Having received childbirth preparation training,
* Absence of a birth attendant in trauma,

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Since pregnancy takes place in the woman's body, it is a woman-oriented study and primiparous women who have completed the gestational period were included in the study.
Enrollment: 44 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Perception of Control and Support in the Birth Scale | 4 months
  The scale was developed by Elizabeth Ford, Susan Ayers and Daniel B. Wright in 2009 under the name Support and Control in Childbirth Scale (SCBS). The Turkish validation of the scale was conducted by Figen İnci, Gözde Gökçe İşbir and Fuat Tanhan in 2015. The scale consists of 33 items and three sub-dimensions: support, control and external control. The sub-dimensions are the health worker's support dimension items 1-12 and the mother's control over her own body and birth sub-dimension items 13-33. The scale is a five-point Likert-type scale as "Strongly Agree", "Agree", "Undecided", "Disagree", "Strongly Disagree". There are 10 negative statements in the scale. The scores that can be obtained from the DCOS scale range from 33 to 165 and these scores were used to determine the level of control and support perceived by women. Cronbach's alpha coefficient of the scale is 0.84. In this study, Cronbach's alpha coefficient was found to be 0.973.

CONTACTS AND LOCATIONS:
Overall Officials: Ayça DEMİR YILDIRIM, PhD, Principal Investigator — Üsküdar University NP Health Campus Institute of Health Sciences Department of Midwifery
Locations (1):
- Uskudar University, Istanbul, Ümraniye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
A research article is planned to make the individual participant data (IPD) available to other researchers.